CLINICAL TRIAL: NCT01281852
Title: A Limited Access Phase I Trial of Paclitaxel, Cisplatin and CTEP Supplied Agent ABT-888 (Veliparib) (NSC#737664) in the Treatment of Advanced, Persistent, or Recurrent Carcinoma of the Cervix
Brief Title: Paclitaxel, Cisplatin, and Veliparib in Treating Patients With Advanced, Persistent, or Recurrent Cervical Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02661; NCI-2011-02661 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GOG-0076HH; CDR0000693745; GOG-0076HH (Other: NRG Oncology); GOG-0076HH (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2011-01-21; First posted 2011-01-24 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Cervical Adenocarcinoma; Cervical Adenosquamous Carcinoma; Cervical Squamous Cell Carcinoma, Not Otherwise Specified; Recurrent Cervical Carcinoma; Stage IVB Cervical Cancer AJCC v6 and v7
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Paclitaxel; Taxes; veliparib

ARMS (1):
- Treatment (paclitaxel, cisplatin, veliparib) (Experimental): Patients receive paclitaxel IV over 3 hours on day 1, cisplatin IV over 1 hour on day 2, and veliparib PO on days 1-7. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cisplatin; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Drug: Veliparib

INTERVENTIONS:
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone''s Chloride; Peyrone''s Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Drug: Veliparib — Given PO
  Other Names: ABT-888; PARP-1 inhibitor ABT-888

SUMMARY:
This phase I clinical trial studies the side effects and best dose of veliparib when given together with paclitaxel and cisplatin and to see how well they work in treating patients with cervical cancer that has spread to other places in the body and usually cannot be cured or controlled with treatment or that has come back. Drugs used in chemotherapy, such as paclitaxel and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Veliparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving more than one drug (combination chemotherapy) and giving chemotherapy together with veliparib may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum-tolerated dose (MTD) and dose-limiting toxicities of ABT-888 (veliparib) when combined with cisplatin and paclitaxel in women with advanced, persistent, or recurrent cervical cancer.

II. To examine the safety of administering ABT-888 when combined with cisplatin and paclitaxel.

III. Once the recommended phase II dose is established, to estimate the efficacy of cisplatin, paclitaxel, and ABT-888 with respect to objective tumor response in patients with advanced, persistent, or recurrent carcinoma of the cervix.

SECONDARY OBJECTIVES:

I. To examine the effects of this regimen on progression-free survival and overall survival.

TERTIARY OBJECTIVES:

I. To determine the proportion of patients with advanced, persistent, or recurrent cancer of the cervix whose tumors demonstrate loss of the Fanconi anemia group D2 (FancD2) foci formation.

III. To determine the association between loss of FancD2 foci formation and progression-free survival, overall survival, and response in this patient population.

OUTLINE: This is a phase I, dose-escalation study of veliparib followed by a phase II study.

Patients receive paclitaxel intravenously (IV) over 3 hours on day 1, cisplatin IV over 1 hour on day 2, and veliparib orally (PO) on days 1-7. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have primary stage IVB, recurrent or persistent squamous cell carcinoma, adenosquamous carcinoma, or adenocarcinoma of the cervix which is not amenable to curative treatment with surgery and/or radiation therapy; histologic documentation of the original primary tumor is required via the pathology report
* All patients in the phase II portion must have measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1; measureable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest dimension to be recorded); each lesion must be >= 10 mm when measured by computed tomography (CT), magnetic resonance imaging (MRI) or caliper measurement by clinical exam; or >= 20 mm when measured by chest x-ray; lymph nodes must be >= 15 mm in short axis when measured by CT or MRI; measurable disease is not required for participation in the phase I portion of this study
* Patients in the phase II portion must have at least one ?target lesion? to be used to assess response on this protocol as defined by RECIST 1.1; tumors within a previously irradiated field will be designated as ?non-target? lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy
* Patients must have a Gynecologic Oncology Group (GOG) Performance Status of 0, 1, or 2
* Recovery from effects of recent surgery, radiotherapy or other therapy

  * Patients should be free of active infection requiring antibiotics (with the exception of uncomplicated urinary tract infection [UTI])
  * Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration; continuation of hormone replacement therapy is permitted
  * At least six weeks must have elapsed from the last administration of chemoradiotherapy, and at least three weeks must have elapsed from the last administration of radiation therapy alone; at least six weeks must have elapsed from the time of any major surgical procedure prior to randomization
* Absolute neutrophil count (ANC) greater than or equal to 1,500/mcl
* Platelets greater than or equal to100,000/mcl
* Hemoglobin >= 9 gm/dL
* Creatinine less than or equal to institutional upper limit normal (ULN) or calculated creatinine clearance (Cockcroft-Gault) >= 60 ml/min
* Calcium, magnesium, phosphate, and potassium levels within institutional normal limits
* Bilirubin less than or equal to 1.5 x ULN
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to 3 x ULN
* Alkaline phosphatase less than or equal to 2.5 x ULN
* Neuropathy (sensory and motor) less than or equal to grade 1
* Patients must have signed an approved informed consent and authorization permitting release of personal health information
* Patients of childbearing potential must have a negative pregnancy test prior to the study entry and be practicing an effective form of contraception; women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* PHASE I: All patients must have received prior chemoradiation
* PHASE I: Patients do not need to have measurable disease

Exclusion Criteria:

* Patients with prior treatment with ABT-888 or other poly adenosine phosphate (ADP) ribose polymerase (PARP) inhibitors
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer and other specific malignancies are excluded if there is any evidence of the other malignancy being present within the last three years; patients are also excluded if their previous cancer treatment contraindicates this protocol therapy
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis OTHER THAN for the treatment of cervical cancer within the last three years are excluded; prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor OTHER THAN for the treatment of cervical cancer within the last three years are excluded; patients may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease
* Patients previously treated with chemotherapy for cervical cancer except when used concurrently with radiation therapy and/or as adjuvant therapy

  * Chemotherapy administered concurrent with primary radiation (e.g., weekly cisplatin) is allowed; adjuvant chemotherapy given following the completion of radiation therapy (or concurrent chemotherapy and radiation therapy) is allowed (e.g., paclitaxel and carboplatin for up to 4 cycles)
* Patients may not be receiving any other investigational agents
* Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to ABT-888 or other agents used in study
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with ABT-888
* Patients with history or evidence upon physical examination of central nervous system (CNS) disease, including primary brain tumor, any brain metastases, or history of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) or subarachnoid hemorrhage within 6 months of the first date of treatment on this study
* Patients who are unable to swallow medication
* Patients who are breast feeding should be excluded

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-03-14 (Actual); Primary Completion 2017-02-11 (Actual); Study Completion 2017-02-11 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicities in the first course of treatment (Phase I) | 21 days
Frequency and severity of adverse effects as assessed by National Cancer Institute Common Terminology Criteria for Adverse Events v. 4.0 | Within 30 days of last protocol treatment
Objective tumor response (complete or partial response) (Phase II) | Up to 5 years

SECONDARY OUTCOMES:
Progression-free survival (Phase II) | From study entry to time of progression or death, whichever occurs first, assessed up to 5 years
Overall survival (Phase II) | From study entry to time of death or the date of last contact, assessed up to 5 years

OTHER OUTCOMES:
Proportion of patients with tumors that demonstrate loss of the FancD2 foci formation | Baseline
  The loss of FancD2 foci formation is associated with progression-free survival, overall survival, and response.

CONTACTS AND LOCATIONS:
Overall Officials: Ritu Salani, Principal Investigator — NRG Oncology
Locations (25):
- United States (25):
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Augusta University Medical Center, Augusta, Georgia
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia

REFERENCES:
- [Derived] Thaker PH, Salani R, Brady WE, Lankes HA, Cohn DE, Mutch DG, Mannel RS, Bell-McGuinn KM, Di Silvestro PA, Jelovac D, Carter JS, Duan W, Resnick KE, Dizon DS, Aghajanian C, Fracasso PM. A phase I trial of paclitaxel, cisplatin, and veliparib in the treatment of persistent or recurrent carcinoma of the cervix: an NRG Oncology Study (NCT#01281852). Ann Oncol. 2017 Mar 1;28(3):505-511. doi: 10.1093/annonc/mdw635. PMID 27998970